CLINICAL TRIAL: NCT07264777
Title: Strategic Daytime Napping Enhances Agility and Lowers Perceived Exertion But Does Not Improve Fatigue Resistance in Adolescent Soccer Players
Brief Title: Strategic Daytime Napping Enhances Agility and Lowers Perceived Exertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate Prof, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PNU-6
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Daytime naps; Anaerobic performance; Fatigue; Exercise physiology; Youth athlete; Agility
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Nap Condition (N0) (Experimental): Participants remained awake during the designated nap period in a quiet, dimly lit environment. No sleep was permitted. Following a 60-minute rest period, agility, repeated-sprint ability, and perceived exertion tests were conducted.
  Interventions: Behavioral: No Nap Condition (N0)
- 25-Minute Nap Condition (N25) (Experimental): Participants took a 25-minute daytime nap opportunity at 14:00 in a dark, quiet room (~22°C). Sleep was verified using Fitbit actigraphy. Sixty minutes after awakening, participants completed agility and repeated-sprint tests with exertion and recovery assessments.
  Interventions: Behavioral: Strategic Napping Protocol
- 45-Minute Nap Condition (N45) (Experimental): Participants took a 45-minute daytime nap opportunity at 14:00 in a dark, quiet room (~22°C). Sleep was verified via Fitbit actigraphy. After a 60-minute post-nap recovery period, agility, repeated-sprint, and perceived exertion measures were collected.
  Interventions: Behavioral: Strategic Napping Protocol

INTERVENTIONS:
Behavioral: Strategic Napping Protocol — This behavioral intervention examines the acute effects of short daytime naps on anaerobic performance and perceived exertion in competitive male soccer players. Each participant completed three nap conditions in a randomized crossover design:
  No Nap (N0): Participants remained awake in a quiet, dimly lit room during the nap opportunity.
  25-Minute Nap (N25): Participants took a 25-minute nap opportunity at 14:00 in a dark, quiet, temperature-controlled room (~22°C).
  45-Minute Nap (N45): Participants took a 45-minute nap opportunity under the same environmental conditions.
  Sleep onset, duration, and wake time were objectively verified using Fitbit Charge 6 actigraphy. To minimize sleep inertia, all performance testing-including the Pro Agility Test, Repeated-Sprint Ability (RSA) Test, and Rate of Perceived Exertion (RPE)-was conducted 60 minutes after awakening.
  Other Names: Controlled Nap Duration Protocol
  Arms: 25-Minute Nap Condition (N25); 45-Minute Nap Condition (N45)
Behavioral: No Nap Condition (N0) — Participants remained awake during the designated nap period in a quiet, dimly lit environment. No sleep was permitted. Following a 60-minute rest period, participants completed the Pro Agility Test and Repeated-Sprint Ability (RSA) Test. Ratings of perceived exertion (RPE) were collected after each sprint to assess subjective effort.
  Arms: No Nap Condition (N0)

SUMMARY:
This study investigates how short daytime naps affect physical performance and perceived exertion in competitive male soccer players. Using a repeated-measures crossover design, sixteen athletes from the U17 and U19 teams of Yeni Malatyaspor completed three experimental sessions separated by 48 hours. Each session involved one of three conditions: no nap (N0), a 25-minute nap (N25), or a 45-minute nap (N45). Participants' agility, repeated-sprint ability, and exertion levels were tested after each condition. Objective sleep data were collected with Fitbit Charge 6 devices, and subjective measures included the Hooper Index, Profile of Mood States, and sleep quality scales.

The study aimed to determine whether strategic napping could acutely improve agility and reduce fatigue during anaerobic performance tasks in soccer players. It was hypothesized that longer naps would enhance agility and lower perceived exertion but would not significantly affect repeated-sprint performance.

DETAILED DESCRIPTION:
repeated-measures crossover design was conducted to examine the acute effects of strategic daytime naps on anaerobic performance in competitive male soccer players. Sixteen players from the Yeni Malatyaspor U17 and U19 teams participated voluntarily. Each participant completed three test sessions under randomized conditions: no nap (N0), 25-minute nap (N25), and 45-minute nap (N45), with a 48-hour recovery period between sessions.

Before testing, all participants underwent familiarization sessions to adapt to nap protocols and performance tests. The nap sessions were held in dark, quiet rooms maintained at ~22°C. Fitbit Charge 6 devices objectively verified nap compliance and duration. Participants abstained from caffeine, alcohol, and strenuous activity for at least 24 hours before testing.

To minimize sleep inertia, physical performance testing began 60 minutes after awakening. The test battery included the Pro Agility Test (to assess change-of-direction speed) and the Repeated-Sprint Ability (RSA) Test (6 × 30 m sprints with 20-second recovery). Heart rate during warm-up and ratings of perceived exertion (RPE) were recorded for standardization and subjective effort assessment.

Subjective measures included the Morningness-Eveningness Questionnaire (MEQ), Hooper Index, Pittsburgh Sleep Quality Index (PSQI), Profile of Mood States (POMS), and Visual Analogue Scales (VAS) for sleep quality and alertness. All players were identified as intermediate chronotypes according to the MEQ.

Anthropometric measurements (height, weight, BMI) were obtained using standardized equipment. Statistical analyses were conducted with SPSS v29, using repeated-measures ANOVA with Bonferroni correction to compare conditions. Effect sizes (ηp², Cohen's dz) and correlations between psychological and performance variables were calculated.

The study hypothesized that short daytime naps would enhance agility and reduce perceived exertion, with longer naps (45 min) providing greater benefits. However, due to the multifactorial nature of repeated-sprint performance, no significant improvements were expected in RSA results. The findings contribute to understanding individualized recovery strategies for soccer players and optimizing nap duration for performance enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Male soccer players aged 16-19 years.
* Active members of the Yeni Malatyaspor U17 or U19 competitive teams.
* In good general health, with no acute or chronic illness or injury.
* Regularly engaged in organized soccer training and competition.
* No habitual daytime napping routine.

Able and willing to comply with all study procedures and testing sessions.

* Obtained informed consent (and parental consent for participants under 18 years).

Exclusion Criteria:

* Current or recent (within 3 months) illness, injury, or infection.
* Diagnosed sleep disorders or reported sleep problems on test days.
* Hyperactivity or other conditions that could interfere with sleep or performance testing.
* Use of medications, caffeine, or substances that could affect sleep or performance.
* Failure to comply with pre-test instructions (e.g., abstaining from strenuous training, alcohol, or caffeine).
* Inability to adhere to nap or testing protocols.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Agility Performance (Pro Agility Test Time) | Measured 60 minutes after awakening in each nap condition (No Nap, 25-min Nap, 45-min Nap).
  Agility performance will be measured using the Pro Agility Test (20-yard shuttle run). The time (in seconds) required to complete the test will be recorded using an electronic timing system (SmarTracks, Germany). Lower times indicate better agility performance.

SECONDARY OUTCOMES:
Change in Repeated-Sprint Ability (RSA) | Measured 60 minutes after awakening in each nap condition.
  Repeated-sprint performance will be assessed using a 6 × 30-meter sprint test with 20-second rest intervals. The total sprint time and mean sprint time will be recorded electronically. Improvements are indicated by reduced sprint times.
Change in Rate of Perceived Exertion (RPE) | Immediately after each nap condition (25-min and 45-min naps).
  Sleep quality and alertness will be assessed using a 10-cm Visual Analogue Scale (VAS). Participants will rate how well they slept and their level of alertness upon awakening. Higher values indicate better subjective sleep quality.
Change in Fatigue, Stress, and Recovery (Hooper Index Scores) | Immediately after completion of each experimental session.
  Description:
  The Hooper Index will be used to assess perceived fatigue, muscle soreness, stress, and sleep quality on a 1-7 Likert scale. Lower scores indicate better recovery and wellness status.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared because the dataset includes identifiable information related to a small group of youth athletes, which could compromise participant confidentiality. Summary results and aggregated findings will be published in scientific journals and shared upon reasonable request.